CLINICAL TRIAL: NCT07208669
Title: Evaluating Whether Treating Elevated Blood Pressure in the Inpatient Setting Impacts Patient Outcomes: the ACT-BP Pilot
Brief Title: Evaluating Whether Treating Elevated Blood Pressure in the Inpatient Setting Impacts Patient Outcomes
Acronym: ACT-BP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Pfoh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Elizabeth Pfoh, Staff/Associate Professor of Medicine, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-1160; 1R34HL173138-01A1 (NIH)
Record Dates: First submitted 2025-09-19; First posted 2025-10-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Blood Pressure Control
Keywords: hypertension; inpatient
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The ACT-BP protocol will be implemented in the intervention units. First, the study team will implement an order on the unit that prompts the nurses to follow the ACT-BP algorithm when a patient has an asymptomatic elevated BP between 160mmHg and 199mmHg. This protocol does not apply to patients who are experiencing hypertensive emergencies or cardiac symptoms. To increase adherence to the ACT-BP protocol, knowledge related to treating the potential underlying causes of an asymptomatically elevated BP and the current state of the evidence will be shared through posters, information sheets and knowledge sessions.
  At the the intervention hospital, the study team will provide caregivers (including physicians) with knowledge related to the state of the evidence for treating asymptomatically elevated BPs through emails, information sheets and one-pagers.
  Interventions: Other: ACT-BP Intervention
- Control Arm (No Intervention): In the control units, care will continue as usual.
  At the the control hospital, caregivers (including physicians) will receive knowledge related to the state of the evidence for treating asymptomatically elevated BPs through an email.

INTERVENTIONS:
Other: ACT-BP Intervention — In our intervention units, the study team will change the unit-based protocols to follow the ACT-BP intervention. First, it prompts the nurse to identify if a patient is experiencing hypertensive emergencies or cardiac symptoms. If so, it suggests calling the physician. If not, it prompts assessment for pain, anxiety, nausea, or hunger and provides evidence-based suggestions. It also prompts monitoring to enhance patients' safety in the case of rapidly rising BP. This algorithm will provide a path for ensuring patients receive appropriate treatment.
  Arms: Intervention Arm

SUMMARY:
The vast majority of the 36.2 million individuals admitted to U.S. hospitals are diagnosed with hypertension and experience an elevated blood pressure (BP) reading during hospitalization. There are no guidelines for managing asymptomatically elevated BPs in the inpatient setting, and growing observational evidence suggests that antihypertensive medication intensification increases harm. The proposed study tests whether a unit-based intervention (ACT-BP) can reduce antihypertensive medication intensification and provides information that is scientifically necessary for designing a cluster-randomized clinical trial that identifies the impact of intensification after experiencing an asymptomatically elevated BP on patient outcomes.

DETAILED DESCRIPTION:
Approximately 50-72% of the 36.2 million individuals admitted to U.S. hospitals are diagnosed with hypertension. Hypertension increases the risk of devastating cardiovascular outcomes, such as strokes, heart attacks, and heart failure. Three-quarters of admitted patients experience at least one elevated blood pressure (BP) (>140/90) during hospitalization. While BP is usually elevated for benign reasons, including pain and anxiety, acutely elevated BP can cause end-organ damage. Currently, no guidelines exist for managing asymptomatically elevated BP in the inpatient setting. There is growing observational evidence that antihypertensive medication intensification for asymptomatically elevated BP can result in adverse outcomes, such as increased readmission. Since observational studies are biased, a large-scale clinical trial is needed to identify whether to treat asymptomatically elevated BPs in the hospital. Yet, it would be unethical and costly to randomize individual patients to receive antihypertensive medication intensification. To overcome these obstacles, this study uses hospital-unit-level intervention, ACT-BP. ACT-BP removes standing orders to call physicians about elevated BPs (which encourages treatment due to social desirability bias), provides education on the potential harm of treating asymptomatically elevated BPs, and suggests alternative procedures (e.g., monitoring BP more frequently). At the end of the study, three specific pieces of knowledge needed to conduct a larger, adequately powered randomized clinical trial will be obtained. First, how much does ACT-BP reduce antihypertensive medication intensification? Second, what refinements will improve its effectiveness? Third, what is the rate of the composite outcome in the intervention and control units?

ELIGIBILITY:
Inclusion Criteria:

* At the unit level: Medical units that do not typically care for patients requiring step-down care.

Exclusion Criteria:

1. Patients less than 18
2. Patients experiencing hypertensive emergencies or cardiac symptoms
3. Patients with active cardiovascular events, such as

   * Stroke
   * Non-ST-elevation
   * Myocardial infarction
   * End-stage renal disease
   * Patients on dialysis
   * Those with acute decompensated heart failure

3. Patients on the unit for more than 10 days

4. Patients transferred in after being in the intensive care unit (ICU)

5. Pregnant and post-partum women

6. Patients discharged within 24 hours of admission

7. Patients whose systolic BP remains below 160 mmHg during hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | From date of first elevated BP reading until the end of hospitalization, assessed up to 13 months.
  The number of new orders for antihypertensive medications or increased doses of an antihypertensive medication for patients who experience an elevated systolic BP (≥160 mmHg and ≤199 mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Pfoh, PhD, MPH, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Cleveland Clinic Hillcrest, Mayfield Heights, Ohio

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the pilot trial will be deposited into a public repository.
Time Frame: At the end of the grant period (August 2027) the supporting information will be available and it will be available for 6 years.
Access Criteria: The research community will have access to our findings at the end of the grant period. Since this is a short (2-year) grant, preliminary results will not be shared. The final dataset of de-identified quantitative results will be shared on Vivli, provided appropriate privacy safeguards are available. Alternatively, the de-identified data will be made available upon request under an FDP Data Use Agreement or similar transfer mechanism. Research can request the qualitative results directly from the Principal Investigator at Cleveland Clinic. Cleveland Clinic will consider each request on an individual basis, with combined input from the Principal Investigator, the Law Department, and the Institutional Review Board. Consistent with Cleveland Clinic policy, the data will be available for six years following the end of the grant period.